CLINICAL TRIAL: NCT01320657
Title: A Randomised Clinical Trial of Orthodontic Treatment With 3 Fixed Appliance Systems Assessed Using Digital Models
Brief Title: A Clinical Trial of Three Fixed Orthodontic Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: East Kent Hospitals University NHS Foundation Trust (Other Government); Southend NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2012-04

CONDITIONS: Orthodontic Treatment
Keywords: Self-ligating; orthodontic; appliance; expansion; dental inclination; Expansion and inclination changes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- InOvation C (Active Comparator): Active Self-ligating Bracket
  Interventions: Device: Conventional orthodontic bracket, passive self-ligating brackets and active self-ligating bracket
- Ovation (Placebo Comparator): Conventional Bracket
  Interventions: Device: Conventional orthodontic bracket, passive self-ligating brackets and active self-ligating bracket
- Damon Q (Experimental): Self-ligating bracket
  Interventions: Device: Conventional orthodontic bracket, passive self-ligating brackets and active self-ligating bracket

INTERVENTIONS:
Device: Conventional orthodontic bracket, passive self-ligating brackets and active self-ligating bracket — Subjects randomized to treatment with one of three fixed orthodontic appliances: Damon Q, InOvation C and Ovation brackets. A pre-determined archwire sequence will be used involving round nickel titanium, rectangular nickel titanium progressing to 0.019 X 0.025 inch stainless steel; specific archwire sequences and appointment intervals will be based on the manufacturer's guidelines. All erupted teeth will have attachments placed from the outset.
  Treated for a minimum of 8 months with the 0.019 X 0.025 inch stainless steel archwire in place for at least 8 weeks.

SUMMARY:
This is a clinical study involving patients undergoing orthodontic treatment with fixed appliances ('train-track braces'). A new type of train-track has recently been marketed. Over 4 million patients worldwide are wearing on of these appliances; this system is considerably more expensive than a normal train-track. However, there is little evidence to support its use.

The effects of three different types of train-track will be assessed with respect to the quality of Orthodontic tooth movement produced. Furthermore, the impact of the different train-tracks on daily life of orthodontic patients will also be measured. Consequently, the investigators will be able to inform orthodontists' decisions relating to the choice of train-track they recommend for their patients. In addition, should the more expensive appliances demonstrate objective or subjective advantage, a significant efficiency saving may develop.

DETAILED DESCRIPTION:
This is a clinical study involving patients undergoing orthodontic treatment with fixed appliances ('train-track braces'). A new type of train-track has recently been marketed. Over 4 million patients worldwide are wearing on of these appliances; this system is considerably more expensive than a normal train-track. However, there is little evidence to support its use.

The effects of three different types of train-track will be assessed in this clinical trial with respect to the quality of Orthodontic tooth movement produced. Furthermore, the impact of the different train-tracks on daily life of orthodontic patients will also be measured. Consequently, the investigators will be able to inform orthodontists' decisions relating to the choice of train-track they recommend for their patients. In addition, should the more expensive appliances demonstrate objective or subjective advantage, a significant efficiency saving may develop.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 16 years and over;
* Fit and well and on no medication;
* In the permanent dentition;
* Undergoing orthodontic treatment in preparation for combined orthodontic-surgical care

or

* Subjects considered suitable for non-extraction maxillary arch treatment if not undergoing combined orthodontic-surgical treatment;
* Crowding less than 6mm

Exclusion Criteria

* Cleft lip and palate and other craniofacial anomalies.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Transverse dimensional changes and bucco-lingual inclination changes | 3 years 10 months
  Width in mm

SECONDARY OUTCOMES:
Subjective pain experience | 3 years 10 months
  Pain score

CONTACTS AND LOCATIONS:
Overall Officials: Robert t Lee, MDS, Principal Investigator — Royal London Dental Institute; Ama Johal, PhD, Study Director — QMUL; Valeria Marinho, PhD, Study Director — QMUL
Locations (2):
- United Kingdom (2):
  - East Kent Hospitals NHS Foundation Trust, Canterbury, Kent
  - Royal London Dental Institute, London

REFERENCES:
- [Derived] Fleming PS, Lee RT, Marinho V, Johal A. Comparison of maxillary arch dimensional changes with passive and active self-ligation and conventional brackets in the permanent dentition: a multicenter, randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):185-93. doi: 10.1016/j.ajodo.2013.03.012. PMID 23910199